CLINICAL TRIAL: NCT05146349
Title: One-Year Impact Evaluation of Minnesota Retaining Employment and Talent After Injury/Illness Network (RETAIN)
Brief Title: Minnesota RETAIN Impact Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Social Security Administration (Unknown); Department of Labor and Industry (Unknown); Minnesota Department of Health (Other Government); Workforce Development, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RTN-MN; OD-32543-18-75-4-27 (Other Grant/Funding Number: SSA)
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-11

CONDITIONS: Any Injury or Illness Acutely Impacting Work
Keywords: RETAIN; Minnesota RETAIN; MN RETAIN; illness recovery; injury recovery; out of work help; work placement assistance; job help; work help; help keeping my job; stay at work; return to work

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RETAIN Programming (Experimental): The experimental group receives the full set of RETAIN intervention activities.
  Interventions: Other: Minnesota RETAIN
- Control (No Intervention): The control group does not receive the full set of RETAIN intervention activities.

INTERVENTIONS:
Other: Minnesota RETAIN — RETAIN projects include a combination of medical provider services, stay-at-work/return-to-work (SAW/RTW) coordination services, and other SAW/RTW services. The evaluation compares the treatment group that is eligible to receive the full set of RETAIN intervention activities and an control group that is not.
  Arms: RETAIN Programming

SUMMARY:
This study is a randomized control trial (RCT) to evaluate the impact of RETAIN program expansion and services on workforce retention and reduction of future workplace disability in the state of MN. Collaboration between partners to implement best practices in early intervention to support injured or ill employees in stay at work and return to work will be implemented.

DETAILED DESCRIPTION:
MN RETAIN is a collaborative program led by the Minnesota Department of Employment and Economic Development (DEED), Minnesota Department of Health (MDH), Department of Labor and Industry (DLI), Mayo Clinic, and Workforce Development Inc (WDI) and includes stakeholders throughout MN.

ELIGIBILITY:
Inclusion Criteria:

* Must have been unable to work for no more than 6 months prior enrollment; 80% of participants must be within 3 months of their last day of work
* 18 years or older
* Minnesota resident
* Works in Minnesota
* Employed or currently in the labor force
* Meets one of the following:

  1. Diagnosis of a work related or personal injury or illness that impacts employment
  2. Invasive procedure (e.g., surgery) within the past 12-weeks or anticipated within the next 8-weeks that impacts employment

Exclusion Criteria:

* Legal representation/litigation at the time of enrollment related to their medical condition.
* Does not have the capacity to give appropriate informed consent
* Employed by a RETAIN healthcare recipient or subrecipient with an existing return to work program for employees (i.e. Mayo Clinic employees)
* Worker's compensation recipients that have a qualified rehabilitation consultant (QRC) or a disability case manager (DCM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Share of enrollees employed in the fourth quarter after enrollment | Measured in the fourth quarter after enrollment
  Share of enrollees employed in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Enrollee earnings in the fourth quarter after enrollment | Measured in the fourth quarter after enrollment
  Sum of enrollee earnings in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Share of enrollees that applied for SSDI or SSI during the 12 months after enrollment | Measured in the 12 months after enrollment
  Share of enrollees that applied for SSDI or SSI during any of the 12 months after enrollment obtained from SSA program data. These files include detailed information about Social Security Disability Insurance (SSDI) and Supplemental Security Income (SSI) applications SSDI and SSI awards, SSDI and SSI benefit amounts and enrollee characteristics (for enrollees who have ever applied for SSA program benefits)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Berk, PhD, Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Mn Retain, Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No